CLINICAL TRIAL: NCT05712681
Title: A Randomized, Open-label, Crossover Phase 1 Clinical Trial to Evaluate Food-Effects on Pharmacokinetics and Pharmacodynamics of Oral Single Dose of JP-1366 Tablet in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate Food-Effects on Pharmacokinetics and Pharmacodynamics of Oral Single Dose of JP-1366 Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JP-1366-105
Record Dates: First submitted 2023-01-13; First posted 2023-02-03 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): T → Washout period(7-14days) → R
  Interventions: Drug: JP-1366 20mg tablet
- Sequence 2 (Experimental): R → Washout period(7-14days) → T
  Interventions: Drug: JP-1366 20mg tablet

INTERVENTIONS:
Drug: JP-1366 20mg tablet — T : JP-1366 20mg tablet after the meal
Drug: JP-1366 20mg tablet — R : JP-1366 20mg tablet under fasting condition

SUMMARY:
To Evaluate Food-Effects on Pharmacokinetics and Pharmacodynamics of Oral single dose of JP-1366 tablet in Healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* A healthy adult aged between 19 and 45 years old
* BMI between 18.0kg/m2 and 27.0kg/m2 at the time of screening

Exclusion Criteria:

* The subject who has clinically significant disease with liver, endocrine system, immune system, nervous system, kidney, cardiovascular disease, mental disorder, the blood of tumor disease, respiratory system or with history of the disease.
* The subject who has a history of gastrointestinal disorders(e.g., gastroesophageal reflux disease, gastrospasm, gastritis, gastrointestinal ulcers, Crohn's disease, etc.) or history of gastrointestinal surgery
* The subject who has an allergic disease(excluding mild allergic rhinitis that does not require administration) or has a history of clinically significant hypersensitivity or adverse reactions to clinical trial drugs or drugs containing the same or other drugs (aspirin, NSAIDs, antibiotics, etc.).
* The subject who has other clinically significant diseases or history
* The subject who has a history of drug abuse
* The subject who cannot withstand the insertion and maintenance of pH catheters

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Cmax of JP-1366 | Pre-dose(0 hour) and up to 34 hours in each period
AUClast of JP-1366 | Pre-dose(0 hour) and up to 34 hours in each period

SECONDARY OUTCOMES:
Gastric pH | Pre-dose(0 hour) up to 24 hours after Investigational product administration

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Central, Seoul, South Korea